CLINICAL TRIAL: NCT03784729
Title: Efficacy of Acupuncture for Intermittent Claudication of Patients With Lumbar Spinal Stenosis
Brief Title: Efficacy of Acupuncture for Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-161-KY
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Spinal Stenosis; Intermittent Claudication
MeSH Terms: conditions — Spinal Stenosis; Intermittent Claudication | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): The acupoints of Shenshu (BL23), "Dachangshu (BL25)", Weizhong (BL40), Chengshan (BL57) and Taixi (KI3) will be inserted.
  Interventions: Other: Acupuncture
- Sham acupuncture (Sham Comparator): The acupoints of Shenshu (BL23), Dachangshu (BL25), Weizhong (BL40), Chengshan (BL57) and Taixi (KI3) will be inserted into a depth of 2-3mm.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — The acupoints of Shenshu (BL23), "Dachangshu (BL25)", Weizhong (BL40), Chengshan (BL57) and Taixi (KI3) will be inserted. For the bilateral" BL25", sterile disposable steel needles (Huatuo, Suzhou, China; 0.3 mm×75 mm) will be inserted to a depth of 50-70mm until until participates feel a sensation similar to electric shock radiating downward to the knees. For the other four acupoints (BL23, BL40, BL57 and KI3), the needles (Huatuo, Suzhou, China; 0.3 mm×40 mm) will be inserted to a depth of 15-25 mm, gently rotated three times and lifted to achieve de qi. It should be noted that the needle at KI3 will be inserted at an angle of 45°obliquely downward. There will be 18 treatment sessions with 3 times a week for continuous 6 weeks and a 30 min treatment per session.
  Arms: Acupuncture
Other: Sham acupuncture — The acupoints of Shenshu (BL23), Dachangshu (BL25), Weizhong (BL40), Chengshan (BL57) and Taixi (KI3) will be inserted into a depth of 2-3mm .No manipulation of needles without deqi will be conducted. The treatment duration and frequency of sessions for participants in the SA group will be the same as in the acupuncture group.
  Arms: Sham acupuncture

SUMMARY:
Degenerative lumbar spinal stenosis (DLSS) is a condition which there is narrowing space of sagittal diameter of spinal canal or nerve root canal for spinal nerve or cauda equina secondary to degenerative changes. DLSS is a common cause of gluteal or lower extremity pain, women and elderly people aged 60-70 are more likely to have DLSS. The early symptoms of this disease are soreness and pain in the low back, gluteal region and posterior region of thighs which can be relieved after resting or changing posture. Being accompanied with gradually aggravated symptoms, patients with DLSS may have neurogenic claudication with hypoesthesia and numbness in lateral lower legs and feet, additionally, few patients may have bowel and bladder disturbances. In accordance of the guidelines of North American Spine Society (NASS), treatment options comprise surgical therapy, epidural steroid injections and physical therapy and transcutaneous electrical stimulation, however, the long-term efficacy of surgery is not superior to that of non-surgical therapy. Moreover, the short-term efficacy of non-surgical therapy is with insufficient evidence. According to a systematic review and recent studies, acupuncture may improve the symptoms of patients and their quality of life, however, there is a lack of placebo-controlled and large sample sized study.

ELIGIBILITY:
Inclusion Criteria:

* Meet the requirements for a clinical diagnosis of DLSS combined with a MRI- or computed tomography (CT)-based radiological diagnosis of central sagittal diameter stenosis of the lumbar spinal canal;
* Have neurogenic intermittent claudication (IC) characterized by progressive pain, numbness, weakness, and tingling of the buttocks and/or legs when standing or walking or with extension of the back, which are relieved upon sitting, lying down, or bending forward [22]; they must always walk in flexion or hunchback posture;
* Have pain of an intensity ≥4 in the buttocks and/or legs when walking, standing, or extending the back, as measured using the Numerical Rating Scale (NRS);
* Have pain in the buttock and/or leg that is more severe than their pain in the lower back;
* Have a Roland-Morris score of at least 7;
* Have received a MRI or CT scan within 1 year that showed the anterior posterior diameter of the canal was ≤12 mm;
* Are aged 50-80 years;
* Have provided signed consent and exhibit willingness to participate in the trial.

Exclusion Criteria:

* Congenital stenosis of the vertebral canal, indications of surgery for DLSS (e.g., segmental muscular atrophy, bowel and bladder disturbances), spinal instability requiring surgery, lumbar tuberculosis, lumbar metastatic carcinoma, or vertebral body/vertebral stenosis segment compression fracture;
* Severe vascular, pulmonary, or coronary artery disease with limited lower extremities motility;
* Clinical comorbidities that could interfere with the collection of data related to pain and walking function such as fibromyalgia, chronic widespread pain, amputation, stroke, Parkinson's disease, spinal cord injury, and dementia;
* Cognitive impairment, such that they are unable to understand the content of the assessment scales or provide accurate data;
* A history of lumbar surgery;
* Plans to become pregnant within 12 months or are already pregnant;
* Received acupuncture treatments for DLSS within the previous 30 days;
* Neurogenic IC mainly manifesting as numbness, weakness, or paraesthesia of the lower extremities instead of pain.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Master, Study Director — Beijing University of Chinese Medicine
Locations (1):
- Guang An Men Hospital, Beijing, China

REFERENCES:
- [Derived] Zhu L, Sun Y, Kang J, Liang J, Su T, Fu W, Zhang W, Dai R, Hou Y, Zhao H, Peng W, Wang W, Zhou J, Jiao R, Sun B, Yan Y, Liu Y, Liu Z. Effect of Acupuncture on Neurogenic Claudication Among Patients With Degenerative Lumbar Spinal Stenosis : A Randomized Clinical Trial. Ann Intern Med. 2024 Aug;177(8):1048-1057. doi: 10.7326/M23-2749. Epub 2024 Jul 2. PMID 38950397
- [Derived] Zhou J, Liu S, Sun Y, Wang W, Liu Z. Efficacy of acupuncture for treatment of intermittent claudication in patients with degenerative lumbar spinal stenosis: protocol for a randomized controlled trial. Trials. 2020 Jul 25;21(1):679. doi: 10.1186/s13063-020-04612-8. PMID 32711555

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture | Sham Acupuncture
Started | 98 | 98
Completed | 86 | 88
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (7.0) | 65.5 (7.8) | 65.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 127
  Male | 36 | 33 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 94 | 95 | 189
  Others | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  China | 98 | 98 | 196
modified Roland-Morris Disability Questionnaire [Mean (Standard Deviation); unit: units on a scale] — RMDQ is the measurement used most widely for back-specific function, and is the fundamental domain of the five standardized core outcomes set for spine disorders. It is modified and validated to assess pain-specific functional status in daily activity experienced by subjects with DLSS by modifying "because of my back" to "because of my back or leg problem". The score of modified RMDQ ranges from 0 (no disability) to 24 (maximum disability), with higher scores indicating greater disability and a reduction of 2 to 3 points as the minimal clinically important difference (MCID).
  units on a scale | 12.6 (3.9) | 12.7 (3.3) | 12.6 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Modified Roland-Morris Disability Questionnaire (RMDQ) Score From Baseline
Description: Modified Roland-Morris Disability Questionnaire (RMDQ) is a reliable pain-specific functional status questionnaire which is easy and simple for patients to complete. The RMDQ includes 24 questions with a score range of 0-24, and there is a phrase "caused by low back pain" after each question which could excluded other reasons for dysfunction of the back. For this scale, higher scores indicate more severe symptoms.
Time Frame: week 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
score on a scale | -4.3 [-5.2 to -3.4] | -3.0 [-3.9 to -2.1]

2. Secondary Outcome: The Change in Modified Roland-Morris Disability Questionnaire (RMDQ) Score From Baseline
Description: as for outcome 1
Time Frame: week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
score on a scale | -4.6 [-5.6 to -3.7] | -2.6 [-3.5 to -1.6]

3. Secondary Outcome: The Change in Modified Roland-Morris Disability Questionnaire (RMDQ) Score From Baseline
Description: as for outcome 1
Time Frame: week 30
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
score on a scale | -4.8 [-5.8 to -3.8] | -3.0 [-4.0 to -2.0]

4. Secondary Outcome: The Percentage of Participants With at Least 30% Reduction From Baseline in the Modified Roland-Morris Disability Questionnaire (RMDQ)
Description: Modified Roland-Morris Disability Questionnaire (RMDQ) is a reliable pain-specific functional status questionnaire including 24 questions with a score range of 0-24. For this scale, higher scores indicate more severe symptoms. The percentage of patients wtih a reduction of at least 30% from baseline in the RMDQ will be calculated.
Time Frame: week 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
percentage of participants | 55.4 [45.0 to 65.8] | 39.5 [29.5 to 49.4]

5. Secondary Outcome: The Percentage of Participants With at Least 30% Reduction From Baseline in the Modified Roland-Morris Disability Questionnaire (RMDQ)
Description: as for outcome 4
Time Frame: week 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
percentage of participants | 65.6 [55.7 to 75.6] | 31.5 [21.7 to 41.2]

6. Secondary Outcome: The Percentage of Participants With at Least 30% Reduction From Baseline in the Modified Roland-Morris Disability Questionnaire (RMDQ)
Description: as for outcome 4
Time Frame: week 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
percentage of participants | 62.5 [52.4 to 72.6] | 44.9 [34.4 to 55.4]

7. Secondary Outcome: The Percentage of Participants With at Least 50% Reduction From Baseline in the Modified Roland-Morris Disability Questionnaire (RMDQ)
Description: Modified Roland-Morris Disability Questionnaire (RMDQ) is a reliable pain-specific functional status questionnaire including 24 questions with a score range of 0-24. For this scale, higher scores indicate more severe symptoms. The percentage of patients wtih a reduction of at least 50% from baseline in the RMDQ will be calculated.
Time Frame: week 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
percentage of participants | 37.9 [27.7 to 48.1] | 25.3 [16.4 to 34.3]

8. Secondary Outcome: The Percentage of Participants With at Least 50% Reduction From Baseline in the Modified Roland-Morris Disability Questionnaire (RMDQ)
Description: as for outcome 7
Time Frame: week 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
percentage of participants | 51.7 [41.2 to 622] | 21.1 [12.6 to 29.8]

9. Secondary Outcome: The Percentage of Participants With at Least 50% Reduction From Baseline in the Modified Roland-Morris Disability Questionnaire (RMDQ)
Description: as for outcome 7
Time Frame: week 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
percentage of participants | 48.3 [37.8 to 58.9] | 27.9 [18.6 to 37.3]

10. Secondary Outcome: Changes in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back as Measured by the Number Rating Scale (NRS) in the Previous 1 Week From Baseline
Description: NRS is a brief scale for assessing pain completed by patients themselves. The scores of NRS ranges from 0 to 10 with 11 grades and higher scores indicates greater pain.
Time Frame: week 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
score on a scale | -2.6 [-3.0 to -2.2] | -1.9 [-2.3 to -1.4]

11. Secondary Outcome: Changes in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back as Measured by the Number Rating Scale (NRS) in the Previous 1 Week From Baseline
Description: as for outcome 10
Time Frame: week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
score on a scale | -3.1 [-3.5 to -2.6] | -1.7 [-2.1 to -1.3]

12. Secondary Outcome: Changes in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back as Measured by the Number Rating Scale (NRS) in the Previous 1 Week From Baseline
Description: as for outcome 10
Time Frame: week 30
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
score on a scale | -3.1 [-3.6 to -2.7] | -1.9 [-2.3 to -1.5]

13. Secondary Outcome: At Least 30% Reductions From Baseline in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back, as Measured by the Number Rating Scale (NRS) for the Previous 1 Week
Description: as for outcome 10
Time Frame: week 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
percentage of participants | 56.1 [45.9 to 66.4] | 41.4 [31.1 to 51.6]

14. Secondary Outcome: At Least 30% Reductions From Baseline in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back, as Measured by the Number Rating Scale (NRS) for the Previous 1 Week
Description: as for outcome 10
Time Frame: week 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
percentage of participants | 69.6 [60.3 to 79.0] | 37.5 [27.3 to 47.8]

15. Secondary Outcome: At Least 30% Reductions From Baseline in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back, as Measured by the Number Rating Scale (NRS) for the Previous 1 Week
Description: as for outcome 10
Time Frame: week 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
percentage of participants | 68.2 [58.6 to 77.8] | 40.9 [30.6 to 51.3]

16. Secondary Outcome: At Least 50% Reductions From Baseline in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back, as Measured by the Number Rating Scale (NRS) for the Previous 1 Week
Description: as for outcome 10
Time Frame: week 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
percentage of participants | 41.1 [30.8 to 51.3] | 24.1 [15.2 to 33.0]

17. Secondary Outcome: At Least 50% Reductions From Baseline in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back, as Measured by the Number Rating Scale (NRS) for the Previous 1 Week
Description: as for outcome 10
Time Frame: week 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
percentage of participants | 57.1 [46.7 to 67.5] | 23.4 [14.5 to 32.3]

18. Secondary Outcome: At Least 50% Reductions From Baseline in the Average Pain Scores for the Buttocks and/or Legs When Walking, Standing, or Extending the Back, as Measured by the Number Rating Scale (NRS) for the Previous 1 Week
Description: as for outcome 10
Time Frame: week 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
percentage of participants | 52.6 [42.1 to 63.1] | 25.0 [15.8 to 34.2]

19. Secondary Outcome: The Changed Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Symptom Severity Domain From Baseline
Description: SSSQ is a short outcome measure for symptoms and functions. SSSQ consists of 18 questions and three domains including symptom severity, physical function, and satisfaction with the degree of treatment. The scores for all three domains are calculated by taking the total score for the domain and dividing it by the number of answered questions, and if more than two items are missing, the scale scores for that domain are considered missing.
  Six questions in the symptom severity domain assess pain of the back, buttocks, legs, or feet as well as pain frequency, numbness, and weakness with scores ranging from 1 to 5, while one question assesses balance with possible scores of 1, 3, and 5. The score of symptom severity domain ranges from 1 to 5, with higher scores indicating worse symptoms.
Time Frame: week 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
score on a scale | -0.7 [-0.8 to -0.6] | -0.5 [-0.7 to -0.4]

20. Secondary Outcome: The Changed Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Symptom Severity Domain From Baseline
Description: as for outcome 19
Time Frame: week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
score on a scale | -0.8 [-0.9 to -0.6] | -0.4 [-0.5 to -0.3]

21. Secondary Outcome: The Changed Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Symptom Severity Domain From Baseline
Description: as for outcome 19
Time Frame: week 30
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
score on a scale | -0.8 [-0.9 to -0.6] | -0.5 [-0.6 to -0.4]

22. Secondary Outcome: The Changed Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Physical Function Domain From Baseline
Description: SSSQ is a short outcome measure for symptoms and functions. SSSQ consists of 18 questions and three domains including symptom severity, physical function, and satisfaction with the degree of treatment. The scores for all three domains are calculated by taking the total score for the domain and dividing it by the number of answered questions, and if more than two items are missing, the scale scores for that domain are considered missing.
  The physical function domain assesses walking distance and ability to walk for pleasure, shopping, and getting around the house or apartment and from the bathroom to the bedroom. This domain has five questions with scores ranging from 1 to 4, and higher scores indicate worse function.
Time Frame: week 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
score on a scale | -0.5 [-0.6 to -0.4] | -0.4 [-0.5 to -0.3]

23. Secondary Outcome: The Changed Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Physical Function Domain From Baseline
Description: as for outcome 22
Time Frame: week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
score on a scale | -0.6 [-0.7 to -0.5] | -0.3 [-0.4 to -0.2]

24. Secondary Outcome: The Changed Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Physical Function Domain From Baseline
Description: as for outcome 22
Time Frame: week 30
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
score on a scale | -0.6 [-0.7 to -0.4] | -0.4 [-0.5 to -0.3]

25. Secondary Outcome: The Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Satisfaction Domain From Baseline
Description: SSSQ is a short outcome measure for symptoms and functions. SSSQ consists of 18 questions and three domains including symptom severity, physical function, and satisfaction with the degree of treatment. The scores for all three domains are calculated by taking the total score for the domain and dividing it by the number of answered questions, and if more than two items are missing, the scale scores for that domain are considered missing.
  The satisfaction domain has four categories (very satisfied, somewhat satisfied, somewhat dissatisfied and very dissatisfied) with a score range of 1 to 4.
Time Frame: week 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
score on a scale | 1.6 [1.5 to 1.8] | 2.1 [1.9 to 2.2]

26. Secondary Outcome: The Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Satisfaction Domain From Baseline
Description: as for outcome 25
Time Frame: week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
score on a scale | 1.7 [1.5 to 1.8] | 2.1 [1.9 to 2.2]

27. Secondary Outcome: The Changed Mean Score of Swiss Spinal Stenosis Questionnaire (SSSQ) in Satisfaction Domain From Baseline
Description: as for outcome 25
Time Frame: week 30
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
score on a scale | 1.7 [1.5 to 1.8] | 2.2 [2.0 to 2.3]

28. Secondary Outcome: The Percentage of Participants With Somewhat Satisfied in the Satisfaction Domain of Swiss Spinal Stenosis Questionnaire (SSSQ)
Description: According to satisfaction domain of the SSSQ, patients scoring 1.5-2.5 points are regarded as somewhat satisfied with the therapy, and those scoring 1.5 points or lower are regarded as very satisfied with the therapy.
Time Frame: week 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
percentage of participants | 48.3 [37.8 to 58.8] | 45.1 [34.5 to 55.3]

29. Secondary Outcome: The Percentage of Participants With Somewhat Satisfied in the Satisfaction Domain of Swiss Spinal Stenosis Questionnaire (SSSQ)
Description: as for outcome 28
Time Frame: week 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
percentage of participants | 41.4 [31.0 to 51.7] | 41.3 [31.1 to 51.5]

30. Secondary Outcome: The Percentage of Participants With Somewhat Satisfied in the Satisfaction Domain of Swiss Spinal Stenosis Questionnaire (SSSQ)
Description: as for outcome 28
Time Frame: week 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
percentage of participants | 45.0 [34.5 to 55.5] | 52.6 [42.2 to 63.0]

31. Secondary Outcome: The Percentage of Participants With Very Satisfied Based on the Satisfaction Domain of Swiss Spinal Stenosis Questionnaire (SSSQ)
Description: as for outcome 28
Time Frame: week 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
percentage of participants | 44.8 [34.3 to 55.3] | 26.4 [17.3 to 35.4]

32. Secondary Outcome: The Percentage of Participants With Very Satisfied Based on the Satisfaction Domain of Swiss Spinal Stenosis Questionnaire (SSSQ)
Description: as for outcome 28
Time Frame: week 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
percentage of participants | 47.1 [36.6 to 57.6] | 26.7 [17.5 to 35.8]

33. Secondary Outcome: The Percentage of Participants With Very Satisfied Based on the Satisfaction Domain of Swiss Spinal Stenosis Questionnaire (SSSQ)
Description: as for outcome 28
Time Frame: week 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
percentage of participants | 47.2 [36.7 to 57.7] | 17.7 [9.7 to 25.7]

34. Secondary Outcome: The Change of Hospital Anxiety and Depression Scale (HADS) Score From Baseline
Description: HADS is validated and standardized for measuring the state of anxiety and depression (0-42, with higher scores indicating severe symptoms). HADS has 2 subscales with 14 items (7 items each), and a total score of 0 to 21 with 0 to 3 for each item.
Time Frame: week 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
score on a scale | -3.8 [-5.0 to -2.6] | -2.7 [-3.8 to -1.5]

35. Secondary Outcome: The Change of Hospital Anxiety and Depression Scale (HADS) Score From Baseline
Description: as for outcome 34
Time Frame: week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 88
score on a scale | -3.1 [-4.3 to -1.8] | -3.0 [-4.3 to -1.7]

36. Secondary Outcome: The Change of Hospital Anxiety and Depression Scale (HADS) Score From Baseline
Description: as for outcome 34
Time Frame: week 30
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 86 | 88
score on a scale | -2.8 [-4.2 to -1.4] | -2.2 [-3.6 to -0.8]

37. Other Pre Specified Outcome: The Percentage of Patients Who Have Expectancy of Acupuncture
Description: Expectancy of acupuncture will be recorded at baseline. Participants will be required to answer two questions: "In general, do you believe acupuncture is effective for treating the illness?" and "Do you think acupuncture will be helpful to improve your symptoms of DLSS?" Participants could choose "Unclear", "Yes" or "No" as the answer.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 98 | 98
Participants
  In general, do you believe acupuncture is effective for treating the illness?: Unclear | 28 | 29
  In general, do you believe acupuncture is effective for treating the illness?: Yes | 65 | 65
  In general, do you believe acupuncture is effective for treating the illness?: No | 5 | 4
  Do you think acupuncture will help to improve your symptoms of lumbar spinal stenosis?: Unclear | 35 | 36
  Do you think acupuncture will help to improve your symptoms of lumbar spinal stenosis?: Yes | 58 | 58
  Do you think acupuncture will help to improve your symptoms of lumbar spinal stenosis?: No | 5 | 4

38. Other Pre Specified Outcome: The Percentage of Patients With Successful Blinding
Description: Patients will be informed that the study involves two types of acupuncture: traditional and modern. Following treatment (sessions 17 or 18) and within 5 minutes, they will be asked: 'Based on your experience, which acupuncture type do you think you received: traditional or modern?' Successful blinding will be defined as the patient indicating they received 'traditional' acupuncture.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 87 | 91
Participants | 76 | 69

39. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Adverse events related to acupuncture include severe pain (assessed by VAS, 7 points at least), broken needle, fainting, local hematoma, localized infection and post-acupuncture discomfortable symptoms such as nausea, vomiting, palpitation, dizziness, headache, anorexia and insomnia, etc. during treatment period. Adverse events irrelevant with the treatment will also be recorded in detail.
Time Frame: week 1 to week 30
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 97 | 98
Participants | 9 | 3

ADVERSE EVENTS:
Time Frame: 31 weeks
Arm/Group | Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 3/98 | 1/98
Other Adverse Events (participants affected / at risk) | 6/98 | 2/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture (N=98) | Sham Acupuncture (N=98)
Lacunar infarction (Nervous system disorders) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Hospitalization to receive surgery (Surgical and medical procedures) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture (N=98) | Sham Acupuncture (N=98)
Subcutaneous hematoma (Skin and subcutaneous tissue disorders) | 1 | 1
Sharp pain (Skin and subcutaneous tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Road traffic accident injury (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT03784729/Prot_SAP_ICF_000.pdf